CLINICAL TRIAL: NCT04088695
Title: Effect of a Web Page Intervention Based on a Motivational Video for Voluntary Blood Donation
Brief Title: Effect of a Web Page Based on a Motivational Video for Voluntary Blood Donation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Peruana Cayetano Heredia (Other)
Responsible Party: Principal Investigator, Yelina Leonor Vásquez Guevara, Researcher, Universidad Peruana Cayetano Heredia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 103851
Record Dates: First submitted 2019-07-11; First posted 2019-09-13 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Blood Donors
Keywords: Blood; Donation; Voluntary

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial conducted online to compare the effect of a web intervention which will be developed through a web page containing a motivational video and an informative text for potential voluntary blood donors. The motivational video or the informative text will be offered randomly to each participant to evaluate the effect of each of them. The website will be offered through social networks Facebook and WhatsApp.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The arm exposed to the intervention video
  Interventions: Other: Video through a web page
- Control (Active Comparator): The control group exposed an informative text.
  Interventions: Other: Informative text

INTERVENTIONS:
Other: Video through a web page — Participants will see a video about blood donation.
  Arms: Intervention
Other: Informative text — Participants will see a brief text about blood donation.
  Arms: Control

SUMMARY:
Voluntary blood donation is currently a key issue in many countries, as the shortage of voluntary donors results in a deficit in the supplies of the Blood Banks of the hospitals. One factor for which there is a low number of voluntary donors is the limited dissemination of information that is given to the population regarding the facilities and benefits of blood donation.

Objective: To evaluate the effect of a web page containing a motivational video and an informative text to promote the voluntary donation of blood disseminated through the use of social networks such as Facebook and WhatsApp.

Design and Participants: Online randomized controlled trial for a group of 102 university students.

Intervention: One group exposed to the intervention with video and the other control group exposed to informative text.

DETAILED DESCRIPTION:
PROBLEM STATEMENT The shortage of voluntary blood donors is a constant worldwide problem, since many lives depend on a transfusion every day to carry out medical or surgical treatment, however, the demand is so high that it exceeds the available number of units of blood. That is why the WHO recommends that at least 2% of the total population donate blood to supply the national demand for blood units. It is known that Peru needs around 520,000 units of blood per year to be able to supply the national demand of blood banks (19). In 2017, only 1.08% of the Peruvian population donated blood.

The shortage of blood supply in the blood banks of hospitals is a problem worldwide. The demand for blood has increased in recent decades. This is because blood and its derivatives are used to attend to procedures that support the patient's well-being. It is due to this high demand that all the countries of the world have found themselves in need of generating national laws and systems that help to boost research and voluntary blood donation.

When developing strategies for the promotion of the voluntrary blood donation, it is necessary to know the perceptions that donors have regarding the donation. A study conducted in a hospital in Lima showed the positive and negative aspects regarding blood donation, which resulted in one of the negative aspects is the limited publicity that is given regarding the blood donation. The donors interviewed suggested that advertising could be done through the internet, spreading the information through emails or through the use of Facebook.

HYPOTHESIS It is proposed that there is a significant difference in the increase in the intention to donate blood voluntarily after exposing the participants to a motivational video about blood donation compared to participants exposed to an informative text about blood donation. Both groups will receive the information (video or text) through a web page.

ELIGIBILITY:
Inclusion Criteria:

* Be between 18 and 30 years old.
* Be a student of the Universidad Peruana Cayetano Heredia.
* Never donated blood

Exclusion Criteria:

-Denial to participate in the study.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Number of participants who were voluntary blood donors after the intervention. | 1 month
  It is desired to know the percentage of participants who will become voluntary blood donors after being exposed to web intervention.

SECONDARY OUTCOMES:
The percentage of the participants intends to donate blood voluntarily after the web intervention. | 1 month
  The percentage of the intention to donate blood in the student population of a private university will be evaluated after being exposed to web intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Yelina L Vasquez, Graduate, Principal Investigator — Universidad Peruana Cayetano Heredia
Locations (1):
- Universidad Peruana Cayetano Heredia, San Martín de Porres, Lima region, Peru

IPD SHARING:
Plan to Share IPD: No